

## CONFIDENTIAL

# STATISTICAL ANALYSIS PLAN

A Phase 3, multicenter, randomized, double-masked clinical trial to assess the efficacy and safety of clobetasol propionate ophthalmic nanoemulsion 0.05% compared to placebo in the treatment of inflammation and pain associated with cataract surgery

## **CLOSE-1 study**

Sponsor Study Code: CLOBOF3-16IA01

**Sponsor** Laboratorios Salvat, S.A.

**Product/Compound/Device** Clobetasol propionate ophthalmic nanoemulsion 0.05%

(SVT-15473)

Phase of the study 3

Author

Company

Address

Telephone number

VersionFinal 3Date09-JUL-2021

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

## **SIGNATURES**

| Sponsor Study Code: | CLOBOF3-16IA01 |
|---|---|
| Author | |
| Name, highest academic level, job title: | |
| Company | |
| Signature: | Date/time: |
| Reviewing Statistician | |
| Name, highest academic level, job title: | |
| Company | |
| Signature: | Date/time: |
| Sponsor Approval | |
| Name, highest academic level, job title: | Enrique Jiménez, MD, Medical Director |
| Company | Laboratorios Salvat, S.A. |
| Signature: | Date/time: |

# Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01

## NCT No.: NCT04246801

## **TABLE OF CONTENTS**

| 1 | INTRODUCTION | 5 |
|---|---|---|
| 2 | STUDY OBJECTIVES | |
| 2.1 | Primary Objective | |
| 2.2 | Secondary Objectives | |
| 3 | ENDPOINTS | |
| 3.1 | Primary Efficacy Endpoint | |
| 3.2 | Secondary Efficacy Endpoints | |
| 3.3 | Secondary Encacy Endpoints | |
| 3.3<br>4 | OVERALL STUDY DESIGN | |
| <del>4</del><br>4.1 | Overview of Study Design | |
| 4.1<br>4.2 | Determination of Sample Size | |
| 4.2<br>5 | DATA SETS TO BE ANALYSED | |
| 5<br>6 | STATISTICAL AND ANALYTICAL PLANS | |
| 6.1 | Changes in the Planned Analyses | |
| 6.2 | Blind Review | |
| 6.2<br>6.3 | Hypotheses and Statistical Methods | |
| 6.3.1 | Definitions | |
| 6.3.2 | Summary Statistics | |
| 6.3.3 | Patient/Patient Data Listings | |
| 6.3.4 | Demographic and Other Baseline Characteristics | |
| 6.3.5 | Primary Efficacy analysis | |
| 6.3.6 | Secondary Efficacy Analyses | . 15 |
| 6.3.6.1 | Key Secondary Efficacy Analysis | |
| 6.3.6.2 | Secondary Analysis | |
| 6.3.7 | Sensitivity Analysis | |
| 6.3.8 | Exposure to Treatment | |
| 6.3.9 | Concomitant Medications | |
| 6.3.10 | Adverse Events | |
| 6.3.11 | Other Safety Assessments | |
| 6.4 | Level of Significance, Multiple Comparisons and Multiplicity | |
| 6.5 | Adjustment for Covariates | |
| 6.6 | Handling of Dropouts and Missing Data | |
| 6.7 | Multicentre Studies | |
| 6.8 | Examination of Subgroups | |
| 6.9 | Interim Analysis | . 22 |
| 6.10 | Reporting Conventions | . 22 |
| 7 | REFERENCES | . 22 |
| 8 | LIST OF OUTPUT | . 23 |
| 8.1 | Tables to be produced for the Clinical Study Report (Section 14 according to IC | СН |
| | E3) | . 23 |
| 8.2 | Listings of individual patient data and other information to be produced for the | |
| | clinical study report (sections 16.1 and 16.2 according to ICH E3) | . 29 |

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01

NCT No.: NCT04246801

#### **ABBREVIATIONS**

ΑE Adverse Event

AESI Adverse Event of Special Interest ATC **Anatomical Therapeutic Chemical** 

**BCVA Best-Corrected Visual Acuity** 

BMI **Body Mass Index** 

CSR Clinical Study Protocol

**eCRF** Electronic Case Report Form

**FAS** Full Analysis Set

**ICH** International Conference on Harmonization

IMP **Investigational Medicinal Product** 

IOP Intraocular Pressure

Medical Dictionary for Regulatory Activities MedDRA

**MMRM** Mixed Model of Repeated Measures **NSAID** Non-Steroidal Anti-Inflammatory Drug

PP Per Protocol PT Preferred Term Q1 25th percentile Q3 75th percentile

QID Four times a day (Quater In Die) REML Restricted Maximum Likelihood

SAE Serious Adverse Event SAF Safety Analysis Set

SAP Statistical Analysis Plan

SOC System Organ Class

STEAE Serious Treatment-Emergent Adverse Event

SUN Standardization of Uveitis Nomenclature

**TEAE** Treatment-Emergent Adverse Event

VAS Visual Analog Scale

**WHO** World Health Organization

Date: 09-JUL-2021

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) is based on Clinical Study Protocol (CSP) Version 2.0 FINAL Amendment 1 dated February 26, 2020.

#### 2 STUDY OBJECTIVES

#### 2.1 Primary Objective

To assess the effect of clobetasol propionate ophthalmic nanoemulsion 0.05% on ocular inflammation associated with cataract surgery after one week of treatment.

## 2.2 Secondary Objectives

#### Key secondary objective

#### Efficacy:

• To assess the effect of clobetasol propionate ophthalmic nanoemulsion 0.05% on eye pain associated with cataract surgery after one week of treatment.

#### Other secondary objectives

#### Efficacy:

- To assess the effect of clobetasol propionate ophthalmic nanoemulsion 0.05% on ocular inflammation associated with cataract surgery
- To assess the effect of clobetasol propionate ophthalmic nanoemulsion 0.05% on eye pain and on eye discomfort associated with cataract surgery

#### Safety:

 To evaluate the safety and tolerability of clobetasol propionate ophthalmic nanoemulsion 0.05%

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

#### 3 **ENDPOINTS**

#### 3.1 **Primary Efficacy Endpoint**

Proportion of patients with anterior chamber cell grade of "0" (absence of cells) compared to placebo at Day 8.

Anterior chamber cell grade will be assessed by the investigator during slit-lamp examination and will be graded on an adapted 6-point scale proposed by the Standardization of Uveitis Nomenclature (SUN) working group (Table 1).

Calla in field\*

Table 1. Grading scheme for anterior chamber cells

<sup>\*</sup>Field size is a 1mm by 1 mm slit beam

| Grade | Cells in field* |
|-------------------------------------------|-----------------|
| 0 | 0 |
| 0.5+ | 1-5 |
| 1+ | 6-15 |
| 2+ | 16-25 |
| 3+ | 26-50 |
| 4+ | >50 |
| *Field size is a dame but dame alik bears | |

#### 3.2 **Secondary Efficacy Endpoints**

#### Key secondary efficacy endpoint

Proportion of patients with VAS pain score of "0" (no eye pain) compared to placebo at Day 8.

Eye pain score will be assessed by the patient before any ocular examination and will be scored by ticking on a continuous scale comprised of a 10 cm horizontal line anchored by two verbal descriptions: "no eye pain" (score of 0) and "worst imaginable eye pain" (score of 10).



The records to be considered are those whose date coincides with the visit to be analyzed for VAS pain score except in model to analyze the change over time in the VAS pain score reported every day compared to placebo.

Proportion of patients with anterior chamber cell grade of "0" compared to placebo at Day 3, Day 15 and Day 29.

Version: Final 3 Study Code: CLOBOF3-16IA01
Date: 09-JUL-2021 NCT No.: NCT04246801

• Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different anterior chamber cell grades.

Sponsor: Laboratorios Salvat, S.A.

- Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different anterior chamber flare grades.
- Proportion of patients with anterior chamber cell grade of "≤0.5+" and flare grade of "0" compared to placebo at Day 3, Day 8, Day 15 and Day 29.
- Proportion of patients with anterior chamber cell grade of "≤1+" compared to placebo at Day 3, Day 8, Day 15 and Day 29.
- Proportion of patients with anterior chamber cell grade of "0" and flare grade of "0" compared to placebo at Day 3, Day 8, Day 15 and Day 29.
- Frequency of different signs of ocular inflammation compared to placebo at Baseline, Day 3, Day 8, Day 15 and Day 29.
- Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different signs of ocular inflammation.
- Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of signs of ocular inflammation.
- Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the visual analog scale (VAS) photophobia score.
- Change from Baseline to Day 8, Day 15 and Day 29 compared to placebo in Snellen bestcorrected visual acuity (BCVA) score.
- Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the VAS pain score.
- Proportion of patients with VAS pain of "0" compared to placebo at Day 3, Day 15 and Day 29.
- Change from baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different discomfort grades.
- Proportion of patients with no discomfort ("None") compared to placebo at Day 3, Day 8, Day 15 and Day 29.
- Change over time in the VAS pain score reported in the patients' diaries compared to placebo.

See previous section 3.1 for anterior chamber cell grade and key secondary efficacy endpoint of this section for eye pain VAS score.

- Anterior chamber cell flare will be assessed by the investigator during slit-lamp examination and will be graded on a 5-point scale proposed by SUN working group.

Table 2. The SUN working group grading scheme for anterior chamber flare

| Grade | Description |
|-------|----------------------------------------|
| 0 | None |
| 1+ | Faint |
| 2+ | Moderate (iris and lens details clear) |
| 3+ | Marked (iris and lens details hazy) |
| 4+ | Intense (fibrin or plastic aqueous) |

Statistical Analysis Plan Sponsor: Laboratorios Salvat, S.A. Version: Final 3 Date: 09-JUL-2021

Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

Signs of ocular inflammation (chemosis, bulbar conjunctival injection, ciliary injection, corneal edema, keratic precipitates) will be assessed by the investigator during slit-lamp examination. Additionally, the severity of these signs of ocular inflammation will be assessed.

Table 3. Signs of ocular inflammation. Chemosis, bulbar conjunctival injection, ciliary injection, corneal edema and keratic precipitates.

| Grade | Description |
|-------|-------------|
| 0 | None |
| 1 | Mild |
| 2 | Moderate |
| 3 | Severe |

Other: The severity of any other sign of ocular inflammation encountered by the investigators (e.g. hypopion, anterior chamber fibrinoid reaction, miosis, papilar or follicular conjunctival reaction, corneal neovascularization) will not be analyzed. They will only be shown in the listings.

- Monocular visual acuity will be completed with the patient's best correction vision in place using the standardized visual acuity measurement **Snellen** Test.
- The eye discomfort will be assessed by using the following categorical scale (Table

Table 4. Eye discomfort

| Grade | Description |
|-------|-------------|
| 0 | None |
| 1 | Mild |
| 2 | Moderate |
| 3 | Severe |

The records to be considered are those whose date coincides with the visit to be analyzed for eye discomfort.

The photophobia VAS is a single-item continuous scale comprised of a 10 cm horizontal line anchored by two verbal descriptors, one for each symptom extreme. For photophobia intensity, the scale is anchored by "no photophobia" (score of 0) and "worst imaginable photophobia" (score of 10 cm). The photophobia VAS is completed by the patient:

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801



The records to be considered are those whose date coincides with the visit to be analyzed for photophobia VAS.

#### 3.3 Secondary Safety Endpoints

- Number, frequency and severity of adverse events (AEs) up to Day 29.
- Number, frequency and severity of serious AEs (SAEs) up to Day 29.
- Proportion of patients discontinuing the study due to AEs.
- Proportion of patients discontinuing the study due to lack of efficacy.
- Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in intraocular pressure (IOP).
- Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in physical and eye examination parameters and vital signs.
- Use of concomitant medications up to Day 29

The IOP will be assessed in both eyes using the Goldmann applanation tonometry method (for details see Appendix 3 of CSP).

#### 4 OVERALL STUDY DESIGN

#### 4.1 Overview of Study Design

This is a Phase 3, randomised, parallel-group, placebo-controlled, double-masked, multicentre study to assess the efficacy and safety of clobetasol propionate ophthalmic nanoemulsion 0.05% in the treatment of inflammation and pain associated with cataract surgery.

All randomized patients will undergo routine cataract surgery according to the investigator's normal procedures being surgery day considered Day -1 of the study, whereas the day of the randomization/first administration will be considered study Day 1. First administration of the Investigational Medicinal Product (IMP) will take place at the study center, whereas the rest of study medication will be dispensed to patients for self-administration at a dosage of one drop every six hours, four times a day (QID) during 14 days as well as a diary to record the drug instillations.

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

Figure 1. Diagram of Study Design



\* Patients who, for any reason, withdraw from the study treatment will be highly encouraged to continue attending all their remaining study visits to collect the most complete efficacy and safety data.

## 4.2 Determination of Sample Size

At least 210 patients from approximately 20 sites in the U.S. will participate in this study. Patients will be randomized in a 2:1 ratio to receive either clobetasol propionate ophthalmic nanoemulsion 0.05 % (N=140) or placebo (N=70) for the treatment of inflammation and pain associated with cataract surgery. Dropouts will not be replaced since the expected dropout rate is low (4%).

The sample size calculation is based on a two group  $\chi 2$  test with a 0.05 two-sided significance level will have 80% power to detect the difference between a proportion with complete resolution of anterior chamber cells in the active group of 0.22 and the placebo group proportion of 0.07 (odds ratio of 3.747) when the sample size is 202.

#### 5 DATA SETS TO BE ANALYSED

The following analysis sets will be used for the statistical analysis and presentation of data:

• Full Analysis Set (FAS): The FAS will be the primary analysis set for the efficacy endpoints and will include all randomized patients. The FAS population will be analyzed according to the planned treatment (rather than treatment actually received).

Statistical Analysis Plan Sponsor: Laboratorios Salvat. S.A. Version: Final 3 Study Code: CLOBOF3-16IA01 Date: 09-JUL-2021

NCT No.: NCT04246801

Full Analysis Set without including rescued subjects (FAS non-RM set): The FAS non-RM will be the analysis set for the efficacy endpoints and will include all randomized patients without including rescued subjects (prohibited medication allowed.

- Safety Analysis (SAF) set The safety set will be the primary analysis set for the safety endpoints and will include all randomized patients who instilled at least one dose of IMP or placebo. The SAF will be analyzed according to the treatment actually received.
- Per Protocol (PP) Population: The PP population set will be tested to confirm the robustness of the efficacy analyses and will include all patients in the FAS who have no major protocol deviations (i.e. patients who comply the protocol sufficiently to ensure that the data exhibits the effects of the IMP or placebo when administered as intended). Protocol violations include: violations of entry criteria, lack of compliance and the use of prohibited medication. The PP population will be analyzed according to the treatment actually received.

Lack of compliance is defined as less than 80% compliance (section 6.3.8).

Efficacy analyses will be based on both the FAS and the PP, but the FAS will be considered the primary analysis population.

Safety analyses will be based on the SAF.

Primary efficacy and key secondary efficacy analysis will be performed for all efficacy endpoints, analyzing:

-all subjects who were randomized (i.e., FAS set),

#### AND

-all subjects who were randomized without including rescued subjects (i.e., FAS non-RM set)

Secondary efficacy analysis will be performed analyzing all subjects included in the FAS non-RM populations, hereinbefore described.

Sensitivity analysis described in the section 6.3.7 will be performed analyzing all subjects included in FAS set populations, hereinbefore described.

For the efficacy endpoints based in PP population (primary efficacy analysis and key secondary at visit 3) will include all patients in the FAS population who have no major protocol deviations. Without violations of eligibility criteria, lack of compliance at visit 3 (see section 6.3.8 for details) and without the use of rescue/prohibited medication until visit 3.

Only study eye will be analysed and presented in tables and the non-study eye will only be included in listings.

#### 6 STATISTICAL AND ANALYTICAL PLANS

The planned tables and listings are presented in Section 8.

#### **Changes in the Planned Analyses** 6.1

The SAP presented in this document will supersede the statistical analysis methods described in the clinical protocol. Any deviations/changes from the planned analyses described in this

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

document will be identified, with justification, in the appropriate section of the clinical study report (CSR).

Any changes in the statistical analyses once the SAP has been finalised and the database has been locked should be documented at clinical study report (CSR).

VAS is one of the most commonly used measures for pain intensity in clinical trials. In the CLOSE-1 study protocol, eye pain experienced by the subjects at Day 8 compared to placebo is defined as the study's key secondary objective.

Pain is considered a personal and highly subjective experience. The essential requisite for valid interpretation and analysis of VAS ratings obtained throughout the study is to ensure reliable and valid assessments of eye pain.

Different studies (Jensen et al., 2003, Aicher et al., 2011) have been performed to establish preliminary consensus on the cut-offs at which VAS pain scores could be considered no pain, mild, moderate, and severe pain.

Aicher and colleagues categorized VAS pain scores as follows: no pain 0-2 mm, mild pain 2-17 mm, moderate pain 17-47 mm, severe pain 47-77 mm, very severe pain 77-96 mm, and most severe imaginable pain 96-100 mm. On the other hand, Jensen and colleagues concluded that any VAS pain score of 0-4 mm tended to be labeled as no pain.

Based on the previous scientific investigations, the below additional secondary objectives shall be analyzed to complete the evaluation of the eye pain assessment currently described in both, the CLOSE- 1 study protocol and the Statistical Analysis Plan.

These additional analyses shall also help to check the consistency of eye pain assessment by means of a continuous variable (0-100 mm VAS) and its analysis from a dichotomic perspective (no pain VAS=0/pain VAS>0) and from the perspective of the continuous variable the eye pain VAS score is.

- (Proportion of patients with VAS pain score of "0-0.2 cm" (no eye pain) compared to placebo at Day 3, Day 8, Day 15 and Day 29)
- (Proportion of patients with VAS pain score of "0-0.4 cm" (no eye pain) compared to placebo at Day 3, Day 8, Day 15 and Day 29)
- In table 14.2.14 both treatment groups (Clobetasol Propinate/Placebo) at each study visit will be compared using t-test or Mann Whitney Wilcoxon test, as applicable for VAS score.

For FAS non-Rescue and FAS populations.

Additional tables to cover these objectives for both populations 14.2.19.1, 14.2.19.2, 14.2.20.1 and 14.2.20.2 will be added.

#### 6.2 Blind Review

A Blind Data Review Meeting (BDRM) is planned to occur before treatment unblinding takes place. The main objective of this meeting is to review data and identify protocol deviations in order to assign patients to all the analysis sets. Details of BDRM will be specified in a separate document.

A review of all major and critical protocol deviations and their potential consequences for the analysis will be conducted during the BDRM. Results and actions taken will be summarized in the Pre-Analysis Review document, which will be finalized before treatment unblinding.

A summary table will be provided including the number of patients with critical and major protocol deviations and the number of clinical and major protocol deviations. The protocol

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

deviations will be listed. The number of patients per study population will be provided. Listings for patients excluded from the SAF, FAS and PP set will be provided.

## 6.3 Hypotheses and Statistical Methods

## 6.3.1 Definitions

| Baseline | ( Visit 1 (Day 1, 24 h after the cataract surgery). |
|---|---|
| Time calculation | Differences between dates to express duration will be calculated as the final date - initial date + 1. To convert these days differences to other units, the following conversion factors will be used: 1 year = 365.25 days and 1 month = 30.4375 days. |
| | Ex. Age = (informed consent date – date of birth + 1) / 365.25 |
| Absolute change | Absolute change from Baseline at Visit X will be calculated as: |
| from Baseline | Absolute change from Baseline = Visit X - Baseline |
| Percentage change | Percentage change from Baseline at Visit X will be calculated as: |
| from Baseline | Percentage change from Baseline [%] = ((Visit X - Baseline)/Baseline) *100 |
| | In case of Baseline = 0 no percentage change from baseline will be calculated. |
| Signs of ocular inflammation (yes/no) | The presence/absence of the different signs of ocular inflammation:<br>Chemosis, Bulbar conjunctival injection, ciliary injection, corneal<br>edema, keratic precipitates will be defined as: |
| | No: grade=0 (absence) |
| | Yes: grade=1, 2 or 3 (presence) |
| Conversion Snellen | Step 1. Mar = Snellen Denominator/Snellen Numerator |
| to LogMar | Step 2. LogMar = log (Mar) |
| | Example: Snellen 20/40 |
| | Mar = 40/20 = 2 |
| | LogMar= log(2) = 0.3 |
| Treatment Emergent<br>Adverse Event | Treatment Emergent Adverse Events (TEAEs) are defined as an event that emerges during treatment having been absent pretreatment or worsens relative to the pre-treatment state: |
| | First dose IMP/Pacebo date ≤ start date AE ≤ last dose IMP/Placebo date |
| Rescue medication | The following prohibited medications will be considered as rescue medication when administered to subjects not responding to IMP or placebo: |
| | <ul> <li>Any systemic or local therapy with corticosteroids (other<br/>than the study drug) or immunosuppressant (except pre-<br/>surgical and/or surgical administration of 1 drop of a topical<br/>NSAID or corticosteroid, at the investigator discretion)</li> </ul> |

Date: 09-JUL-2021

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01

NCT No.: NCT04246801

| | <ul> <li>Any topical ocular medication (except preservative-free antibiotics for prophylactic purposes and preservative-free artificial tears)</li> <li>Any systemic NSAID or opioids drugs (except occasional use of OTC formulations titrated no more than one single dose per week)</li> </ul> |
|---|---|
| Relative day | The relative day of an event that occurs prior to administration of IMP: |
| | Relative day = (Start date)-(Date of administration of IMP). |
| | The relative day of an event that occurs on the same day or after administration of IMP: |
| | <ul> <li>Relative day = (Start date)-(Date of administration of<br/>IMP)+1.</li> </ul> |
| | Consequently, Day 1 is the same day as the day of administration of IMP, Day -1 is the day before, and Day 2 is the day after. |

## 6.3.2 Summary Statistics

Data will be summarised by means of summary statistics. For continuous data the following summary statistics will be presented: number of observations, mean, standard deviation (SD), minimum, Q1, median, Q3 and maximum. 95% CI of the mean will also be presented for efficacy and safety data. Change from baseline to each post-baseline visit will be also described using descriptive statistics. Categorical data will be presented as counts and percentages.

Summary statistics will be presented by treatment group and visit, as applicable.

Certain presentations (withdrawals, patient exclusion from datasets, baseline and background characteristics and primary efficacy data) may be broken down by study center, if relevant.

All data collected during study follow-up will be displayed and analyzed according to the actual visit data in the eCRF.

#### 6.3.3 Patient/Patient Data Listings

Data collected in the eCRF will generally be listed. eCRF check questions and reminders will not be listed.

Listings will be sorted by study center, patient number, visit (where applicable) and time point (where applicable).

All derived data will be presented in the corresponding data listings.

#### 6.3.4 Demographic and Other Baseline Characteristics

Patient disposition, demographic data and other baseline data will be listed and presented using summary statistics.

Demographic data:

Date: 09-JUL-2021

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

Age, gender, ethnicity, race, weight (pounds), height (inches) and BMI will be summarized by treatment regimen and overall. SAF, FAS and PP population will be used for this presentation.

#### Relevant Medical History:

Medical history data will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA), the latest versionMedical history will be summarized for the SAF by treatment regimen and overall on a per-patient basis (e.g., if a patient reported the same event repeatedly the event will be counted only once at the specific level of display). Absolute counts (n) and percentages (%) will be presented for the number of patients with at least one Medical History event, and per System Organ Class (SOC) and per Preferred Term (PT) within SOC.

A listing will present all history-related data for the SAF.

#### Other clinical baseline characteristics:

Urine pregnancy test results and cataract diagnosis date and study eye will be listed for the SAF. Patient disposition will be presented, based on individual study examination dates and end of study status. A listing will be provided (if applicable) for discontinued patients.

#### 6.3.5 Primary Efficacy analysis

The primary efficacy endpoint in this clinical trial is the proportion of patients with anterior chamber cell grade of "0" (absence of cells) compared to placebo at Day 8.

The statistical hypothesis that will be tested for primary efficacy is described as:

- Null Hypothesis ( $H_0$ ): The difference in proportion of patients with anterior chamber cell grade of "0" at Day 8 between treatment regimes = 0.
- Alternative Hypothesis (H₁): The difference in proportion of patients with anterior chamber cell grade of "0" at Day 8 between treatment regimes ≠ 0.

The aim of the primary analysis of this study is to assess the superiority of clobetasol propionate ophthalmic nanoemulsion 0.05% compared to placebo with respect to the primary efficacy endpoint. The primary analysis will be based on a single study eye for each patient. Each patient's study eye will be defined as the surgery eye.

A Chi-Square test will be employed to test the proportion of study eyes with complete clearing of anterior chamber cells (count cell = 0) at Visit 3 (Day 8  $\pm$  1 day) without receiving rescue medication as compared between clobetasol propionate ophthalmic nanoemulsion 0.05% dosed QID and placebo dosed QID. The proportion of eyes with absence of cells (anterior chamber cell grade=0) together with its 95% confidence interval (CI) will be presented. Analysis will be conducted both in FAS and PP to test the robustness of the results.

#### 6.3.6 Secondary Efficacy Analyses

#### 6.3.6.1 Key Secondary Efficacy Analysis

The key secondary efficacy endpoint is the proportion of patients with VAS pain score of "0" (no eye pain) compared to placebo at Day 8.

The key secondary analysis will be based on a single study eye for each patient. Each patient's study eye will be defined as the surgery eye.

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01

NCT No.: NCT04246801

A Chi-Square test will be performed to test the proportion of study eyes with no pain (VAS = 0) at Visit 3 (Day 8 ± 1 day) without receiving rescue medication as compared between clobetasol propionate ophthalmic nanoemulsion 0.05% dosed QID and placebo dosed QID. The proportion of eyes with no pain together with its 95% confidence interval (CI) will be presented.

Analysis will be conducted both in FAS and PP to test the robustness of the results.

## 6.3.6.2 Secondary Analysis

The secondary efficacy endpoints are described in Section 3.2. All secondary efficacy endpoints defined in this section will be analysed as exploratory.

For categorical variables, a summary of these endpoints will be presented at each specified timepoint by treatment group and will include the number and percentage of each category with the 95% CI. A chi-square test or Fisher Exact test, as appropriate will be performed to compare proportions between treatments at each timepoint.

For continuous variables: VAS photophia, Snellen best-corrected visual acuity (BCVA) score and VAS pain score, a summary of these endpoints will be presented at each specified timepoint by treatment group. Change from baseline will be derived and presented in the same way.

For variables: Anterior chamber cell grades, anterior chamber flare grades, severity of signs of ocular inflammation and eye discomfort grades categorical and continuous summary statistics will be presented, changes from baseline will also be derived and will be presented as increase, decrease or not change table. In the same way, a table with 2 categories: Improvement and no improvement (increase+no change) will be presented. A chi-square test or Fisher Exact test will be performed to compare proportions between treatments:

| Change from baseline to Day 3 | | |
|-------------------------------|---------|---------|
| Anterior Chamber Cell Grade | IMP | Placebo |
| Decrease (Improvement) | n (%) | n (%) |
| No change | n (%) | n (%) |
| Increase (Worsening) | n (%) | n (%) |
| P value chi-square or Fisher | p-value | |
| Improvement | n (%) | n (%) |
| No Improvement | n (%) | n (%) |
| | p-v | /alue |

No Improvement = increase + no change

For the variables mentioned above, to see the proportion of patients with different grades, a descriptive table like the following will also be built, no statistical inference will be made:

| Grade | IMP | | | Placebo | | |
|-------|----------|-------|--------|----------|-------|--------|
| Grade | Baseline | Day X | Change | Baseline | Day X | Change |
| 0 | n (%) | n (%) | (%) | n (%) | n (%) | (%) |

Date: |09-JUL-2021|

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

| 0.5+ | n (%) | n (%) | (%) | n (%) | n (%) | (%) |
|------|-------|-------|-----|-------|-------|-----|
| 1+ | n (%) | n (%) | (%) | n (%) | n (%) | (%) |
| 2+ | n (%) | n (%) | (%) | n (%) | n (%) | (%) |
| 3+ | n (%) | n (%) | (%) | n (%) | n (%) | (%) |
| 4+ | n (%) | n (%) | (%) | n (%) | n (%) | (%) |

Between treatment comparison of the evolution over time will be analysed using a Restricted Maximum Likelihood (REML)-based repeated measures approach (Mixed Model Repeated Measures [MMRM]). The model for analysis will include the change from baseline as a dependent variable, the baseline score as a cavariate, the categorical fixed effects of treatment (IMP, Placebo) and visit and the interaction treatment\*visit. An unstructured (co)variance structure will be used to model the within-patient errors. If this analysis fails to converge, alternative covariance structures will be tested. Akaike's information criterion will be used to determine the best fit (smaller AIC).

If it is not possible to apply a MMRM due to the non-normality of the variable, the Mann Whitney Wilcoxon test will be performed.

Secondary efficacy analyses will be performed on the FAS population.

The PP population set will be also tested to confirm the robustness of the secondary analyses.

#### 6.3.7 Sensitivity Analysis

Sensitivity analysis will be carried out for possible intercurrent events such as discontinuation due to AE, lack of efficacy and use of rescue and prohibited medication. New estimands associated to each intercurrent event will be added to the already existing primary estimand accordingly.

#### 6.3.8 Exposure to Treatment

Subjects will record each IMP or placebo administration (e.g., one drop every six hours, during 14 days) on their dispensed diaries.

Compliance is defined as the percentage of actual doses the patient instilled with respect to the number of total doses planned. The planned dose is always one drop of IMP or placebo. Compliance will be summarized categorically (<80%, ≥80% and 100%) by treatment regime. It will be calculated as follows:

Compliance of IMP/Placebo administered %= (num. of doses instilled / num. of planned doses) )(ml))\*100

#### Planned doses=56

Compliance at last visit with IMP/Placebo is defined as the percentage of actual doses the patient instilled with respect to the number of total doses planned at the time of the last visit with IMP/Placebo.

Compliance of IMP/Placebo administered % at last visit with IMP/Placebo = (num. of doses instilled / num. of planned doses at last visit with IMP/Placebo))(ml))\*100

Date: 09-JUL-2021 NCT No.: NCT04246801

Planned doses at last visit with IMP/Placebo = (End date IMP/Placebo exposure – First date IMP/Placebo exposure+1)\*4.

Sponsor: Laboratorios Salvat, S.A.

Study Code: CLOBOF3-16IA01

Compliance at visit 3 (day 8±1) is defined as the percentage of actual doses the patient instilled with respect to the number of total doses planned at visit 3.

Compliance of IMP/Placebo administered % at visit 3= (num. of doses instilled / num. of planned doses at visit 3) (ml))\*100

#### Planned doses at visit 3=32

In case a scheduled dose was not administered (missed) the missed dose and the reason will be captured in the eCRF as per the patient diary and tabulated by treatment regimen.

All compliance data will be summarized and listed for the SAF.

#### 6.3.9 Concomitant Medications

All concomitant medications/therapies will be classified according to ATC level 3 group text and generic medication name. The medications will be divided into two categories based on start date and end date: Prior Medications and Concomitant Medications: .

- Prior Medications: start date and end date before first day of IMP
- Concomitant Medications:
  - Start date before first day of IMP and end date after or on same day as first day of IMP or no end date, i.e. ongoing after first day of IMP; or
  - Start date after or on same day as first day of IMP

Within concomitant medications, a distinction will be made between rescue medication and prohibited medication.

Incomplete dates will be handled as follows:

- If the start and stop date for a concomitant medication are completely missing, it will be assumed that the medication was started before treatment and classified as Prior Medication.
- If only the start date is missing the medication will be classified as:
  - o Prior if end date is before first day of IMP
  - Concomitant if end date is on or after first day of IMP
- If only the end date is missing the medication will be classified as
  - Concomitant if start date is before or on same day as Day 15
- If the year and/or month are available, medication start in relation to the first day of IMP will be evaluated as close as possible (e.g., if only the year when the medication was started is available and ongoing is checked, the medication will be classified as a Concomitant Medication).
- If the medication was started in the same month as the first day of IMP, the medication will be classified as a Concomitant Medication.

Relative day will generally be calculated for all medications except for the ones with an incomplete start date.

Data will be listed for the SAF. Subject's medications will be presented separately for each timing (i.e. prior, and concomitant medications) in 2 summary tables. In addition, a summary table for rescue and prohibited medication will be presented distinguishing each one in a column.

Study Code: CLOBOF3-16IA01 Date: 09-JUL-2021 NCT No.: NCT04246801

In the listings will show whether the concomitant medication is rescue medication or prohibited medication.

Sponsor: Laboratorios Salvat, S.A.

Rescue medication shall be as reported as such in the eCRD. The following ATC3 codes of concomitant medication will be considered as prohibited medication if they are not classified as rescue medication (all medications will be reviewed and it will be considered whether any medication should be included or excluded in the prohibited classification):

- D07A Corticosteroids, plain
- D07B Corticosteroids, combinations with antiseptics
- D07C Corticosteroids, combinations with antibiotics
- D07X Corticosteroids, other combinations
- G01B Combinations of corticosteroids and antiinfectives for gynaecological use
- A01AC Corticosteroids for local oral treatment
- D01A Corticosteroids in combination with antifungals
- D10AA Corticosteroids, combinations for treatment of acne
- C05AA Antihemorrhoidals with corticosteroids
- S01B Antiinflammatory agents
- S02B Corticosteroids
- S02C Corticosteroids and antiinfectives in combination
- S03B Corticosteroids
- S03C Corticosteroids and antiinfectives in combination.
- H02 Corticosteroids for systemic use.
- L04A Immunosuppressants
- M01A Antiinflammatory and antirheumatic product, non-steroids
- N02BE NSAIDs in combination with paracetamol.
- M01B Salicylates in combination with corticosteroids.
- M01B Combinations of antiinflammatory/antirheumatic agents
- N02A Opioids
- Any ATC3 with ocular route except for S01A, S03A (Antiinfectives) preservative-free for prophylactic purposes and S01X (Other ophthalmologicals) preservative-free.

#### 6.3.10 Adverse Events

AEs data are collected on the 'Adverse Events' eCRF form.

AEs will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) system, the latest version and tabulated by System Organ Class (SOC) and by Preferred Term (PT).

A Treatment-Emergent Adverse Event (TEAE) is defined as an AE observed after starting administration of IMP or placebo (see Section 6.3.1).

TEAEs will be summarized by presenting, for each treatment regimen, the number of events and the number and percentage of patients with:

Study Code: CLOBOF3-16IA01 Date: 09-JUL-2021 NCT No.: NCT04246801

Sponsor: Laboratorios Salvat, S.A.

- Any TEAE
- Any Serious Treatment Emergent Adverse Event (STEAE)
- Any TEAE of Special Interest (TEAESI)
- Any TEAE related to IMP/Placebo
- Any TEAE leading to treatment discontinuation (drug withdrawn)
- Any STEAE related to IMP/Placebo
- Any TEAESI related to IMP/Placebo

The number and percentage of TEAEs by causality and the number and percentage of mild moderate and severe TEAEs will be tabulated by SOC, PT and treatment arm. All tables with TEAEs by SOC and PT stratified by treatment regimen will only be counted by patient once within each PT.

The following tables will be provided with TEAEs by SOC and PT stratified by treatment regimen: TEAEs, TEAEs related to IMP/Placebo, TEAEs leading to discontinuation, STEAEs, STEAEs related to IMP/Placebo, TEAESI and TEAESIs related to IMP/Placebo.

TEAEs, STEAEs and TEAESIs will be tabulated by severity (mild, moderate or severe) and relationship to treatment (No: not related, unlikely related, Yes: possible, probable and certain). If a patient has more than one event with the same PT, the AE will only be counted once and the worst/maximal severity and the worst/strongest relationship will be used.

A listing of all AEs will be presented, whether treatment emergent or not. TEAEs will be flagged in this listing. A separate listing for deaths, STEAEs, AESIs and TEAEs leading to discontinuation will be provided (if any).

The following AEs (SOC, PT) of special interest (AESI) will be evaluated by Investigators at all study visits and time points (as applicable):

- IOP rise over 30 mmHg (SOC- INVESTIGATIONS, PT-INTRAOCULAR PRESSURE INCREASED)
- Pain/discomfort associated with IMP instillation (SOC-EYE DISORDERS, PT-EYE PAIN, OCULAR DISCOMFORT and related with IMP)

Additionally, a descriptive table (14.3.1.2.2) of ocular adverse events will be presented by SOC and PT.

SAF will be used for all AE related summaries.

As stated in the study protocol, treatment arms will be compared with respect to safety endpoints descriptively only. No further inferential comparison will be carried out.

#### 6.3.11 Other Safety Assessments

#### Physical Examination

Full physical examination will consist of assessment of head, eyes, ears, nose throat, mouth, cardiovascular, respiratory, digestive, urogenital, musculoskeletal, nervous/psycological, endocrine/metabolic, hematologic, dermatological, allergies, inmunological and other. The observed values for the physical examination will be recorded in the eCRF by the investigator as "normal" or "abnormal" and if abnormal, assessed as "clinically significant" or "not clinically significant".

The Investigator will perform full physical examinations at the Screening visit and at the Early Termination visit.

Date: 09-JUL-2021

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

The investigator will perform physical examination following the usual standards of patients' examination at each study site.

#### **Eye Examination**

Pupil function, ocular alignment and motility, visual field by confrontation test, and anterior vitreous will be assessed for normality and clinically significance at the Screening visit and at the Early Termination visits.

#### Vital Signs

Vital signs will be assessed 15 minutes before any ocular assessment and at least 30±10 minutes before the first study medication administration. For all vital signs parameters (systolic and diastolic blood pressure, heart rate and body temperature) summary statistics will be produced for observed values by visit.

Vital signs data will be listed by patient. All clinically significant abnormal values will be flagged in this listing.

#### Indirect Ophthalmoscopy

Vitreous humor, central retina, peripheral retina, optic nerve disc and retinal vasculature will be assessed for normality and clinically significance at the Screening, Baseline, Visit 4, Visit 5 and at the Early Termination visit.

Outputs will be based on the SAF.

#### 6.4 Level of Significance, Multiple Comparisons and Multiplicity

All statistical hypotheses will be two-sided and will be performed using a 5% significance level. No adjustment for multiple comparisons or corrections for multiplicity are foreseen.

#### 6.5 Adjustment for Covariates

Baseline value will be used as a covariate in the MMRM analyses for the continuous secondary efficacy endpoints (see Section 6.3.6).

#### 6.6 Handling of Dropouts and Missing Data

No missing imputation methods are foreseen. As described in the CSP, any missing, unused, or spurious data will be noted in the final Clinical Study Report (CSR) and presented in the data listings.

In all listings, missing or incomplete dates should be left as they have been recorded. However, for calculation / sorting / assignation based on dates, the following method will be used, in the event that any date is incomplete after Data Management processing and this date needs to be used for calculation:

- if no field is available: no imputation will be performed,
- if only the year is available: Day "01" and month of "July" will be imputed,
- if the month and year are available: Day "15" will be imputed.

Date: 09-JUL-2021 NCT No.: NCT04246801

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01

#### 6.7 Multicentre Studies

As stated in the CSP, none of the analyses will be adjusted by study center.

#### 6.8 Examination of Subgroups

NA

#### 6.9 Interim Analysis

No formal Interim Analysis is foreseen for this study.

## 6.10 Reporting Conventions

P-values ≥0.0001 will be reported to four (4) decimal places; p-values less than 0.0001 will be reported as <0.0001. The mean and median will be displayed to one decimal place greater than the original value and the measure of variability (e.g., standard deviation) will be displayed to two decimal places greater than the original value.

#### 7 REFERENCES

- 1- ICH E9 Statistical principles for clinical trials (definition Treatment Emergent An event that emerges during treatment having been absent pre-treatment, or worsens relative)
- 2- Jensen et al., 2003. Interpretation of Visual Analog Scale Ratings and Change Scores: A Reanlaysis of Two Clinical Trials of Postoperative Pain.
- 3- Aicher et al., 2011. Pain measurement: Visual Analogue Scale (VAS) and Verbal Rating Scale (VRS) in clinical trials with OTC analgesics in headache.

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 Date: 09-JUL-2021 NCT No.: NCT04246801

#### 8 LIST OF OUTPUT

#### 8.1 Tables to be produced for the Clinical Study Report (Section 14 according to ICH E3)

Demographic data and baseline characteristics will be showed stratifying by treatment group (IMP and placebo) and overall.

Efficacy and safety analysis tables will be showed stratifying by treatment group, as well as each timepoint, as applicable.

For continuous variables, summary statistics will be included in the MMRM tables.

## 14.1 DEMOGRAPHIC DATA

#### Patient disposition

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.1.1 | Patient disposition: Number of patients in each analysis set and reason for exclusion | ALL | Х |
| 14.1.2 | Number of patients by visit | ALL | |
| 14.1.3 | Reason for finish the study prematurely | ALL | |

#### **Demographic and baseline characteristics**

| Table | Title | Pop | Top.Line |
|--------|--------------------------|-----|----------|
| 14.1.4 | Demographics | SAF | |
| 14.1.5 | Urine pregnancy test | SAF | |
| 14.1.6 | Cataract diagnosis | SAF | |
| 14.1.7 | Relevant Medical History | SAF | |

#### 14.2 EFFICACY DATA

## **Primary efficacy analysis**

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.2.1.1 | Percentage of patients with anterior chamber cell grade of "0" compared to placebo at Day 8 | FAS | X |
| 14.2.1.2 | Percentage of patients with anterior chamber cell grade of "0" compared to placebo at Day 8 | PP at<br>Visit 3 | |
| 14.2.1.3 | Percentage of patients with anterior chamber cell grade of "0" compared to placebo at Day 8 | FAS<br>non-<br>RM | Х |

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

# Main Secondary efficacy analysis

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.2.2.1 | Proportion of patients with VAS pain score of "0" (no eye pain) compared to placebo at Day 8. | FAS | X |
| 14.2.2.2 | Proportion of patients with VAS pain score of "0" (no eye pain) compared to placebo at Day 8. | PP at<br>Visit 3 | |
| 14.2.2.3 | Proportion of patients with VAS pain score of "0" (no eye pain) compared to placebo at Day 8. | FAS<br>non-<br>RM | X |

# Secondary efficacy analysis

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.2.3.1 | Proportion of patients with anterior chamber cell grade of "0" compared to placebo at Day 3, Day 15 and Day 29 | FAS<br>non-<br>RM | X |
| 14.2.3.2 | Proportion of patients with anterior chamber cell grade of "0" compared to placebo at Day 3, Day 15 and Day 29 | FAS | |
| 14.2.3.3 | Proportion of patients with VAS pain score of "0" (no eye pain) compared to placebo at Day 3, Day 15 and Day 29. | FAS<br>non-<br>RM | X |
| 14.2.3.4 | Proportion of patients with VAS pain of "0" compared to placebo at Day 3, Day 15 and Day 29. | FAS | |
| 14.2.4.1 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different anterior chamber cell grades. Improvement and no Improvement table. | FAS<br>non-<br>RM | |
| 14.2.4.2 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different anterior chamber cell grades. Descriptive table | FAS<br>non-<br>RM | |
| 14.2.5.1 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different anterior chamber flare grades. Improvement and no Improvement table. | FAS<br>non-<br>RM | |
| 14.2.5.2 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with different anterior chamber flare grades. Descriptive table | FAS<br>non-<br>RM | |
| 14.2.6. | Proportion of patients with anterior chamber cell grade of "≤0.5+" and flare grade of "0" compared to placebo at Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM | |
| 14.2.7. | Proportion of patients with anterior chamber cell grade of "≤1+" compared to placebo at Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM | |

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

| 14.2.8. | Proportion of patients with anterior chamber cell grade of "0" and flare grade of "0" compared to placebo at Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM |
|---|---|---|
| 14.2.9.1 | Frequency of chemosis (yes/no) compared to placebo at Baseline, Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM |
| 14.2.9.2 | Frequency of bulbar conjunctival injection (yes/no) compared to placebo at Baseline, Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM |
| 14.2.9.3 | Frequency of ciliary injection (yes/no) compared to placebo at Baseline, Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM |
| 14.2.9.4 | Frequency of corneal edema (yes/no) compared to placebo at Baseline, Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM |
| 14.2.9.5 | Frequency of keratic precipitates (yes/no) compared to placebo at Baseline, Day 3, Day 8, Day 15 and Day 29. | FAS<br>non-<br>RM |
| 14.2.10.1 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with chemosis (yes/no) | FAS<br>non-<br>RM |
| 14.2.10.2 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with bulbar conjunctival injection (yes/no) | FAS<br>non-<br>RM |
| 14.2.10.3 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with ciliary injection (yes/no) | FAS<br>non-<br>RM |
| 14.2.10.4 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with corneal edema (yes/no) | FAS<br>non-<br>RM |
| 14.2.10.5 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the proportion of patients with keratic precipitates (yes/no) | FAS<br>non-<br>RM |
| 14.2.11.1 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of chemosis. Improvement or no Improvement. | FAS<br>non-<br>RM |
| 14.2.11.2 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of chemosis. Descriptive table | FAS<br>non-<br>RM |
| 14.2.11.3 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of bulbar conjunctival injection. Improvement or no Improvement. | FAS<br>non-<br>RM |
| 14.2.11.4 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of bulbar conjunctival injection. Descriptive table | FAS<br>non-<br>RM |

Improvement

14.2.15.2

14.2.16.1

14.2.16.2

14.2.17

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

| 14.2.11.5 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of ciliary injection. Improvement or no Improvement | FAS<br>non-<br>RM | |
|---|---|---|---|
| 14.2.11.6 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of ciliary injection. Descriptive table | FAS<br>non-<br>RM | |
| 14.2.11.7 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of corneal edema. Improvement or no Improvement. | FAS<br>non-<br>RM | |
| 14.2.11.8 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of corneal edema. Descriptive table | FAS<br>non-<br>RM | |
| 14.2.11.9 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of keratic precipitates. Improvement or no Improvement | FAS<br>non-<br>RM | |
| 14.2.11.10 | Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the severity of keratic precipitates. Descriptive table | FAS<br>non-<br>RM | |
| 14.2.12 | MMRM. Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the visual analog scale (VAS) photophobia score. | FAS<br>non-<br>RM | |
| 14.2.13 | MMRM. Change from Baseline to Day 8, Day 15 and Day 29 compared to placebo in Snellen best.corrected visual acuity (BCVA) score. | FAS<br>non-<br>RM | |
| 14.2.14 | MMRM. Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in the VAS pain score. | FAS<br>non-<br>RM | X |
| 14.2.15.1 | Change from baseline to Day 3, Day 8, Day 15 and Day 29 | FAS | |

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

| 14.2.18 | Percentage of patients with anterior chamber cell grade of "0" compared to placebo at Day 8. Sensitivity Analysis | FAS<br>non-<br>RM | |
|---|---|---|---|
| 14.2.19.1 | Proportion of patients with VAS pain score of "0-0.2 cm" (no eye pain) compared to placebo at Day 3, Day 8, Day 15 and Day 29 (FAS non-RM set). | FAS<br>non-<br>RM | X |
| 14.2.19.2 | Proportion of patients with VAS pain score of "0-0.2 cm" (no eye pain) compared to placebo at Day 3, Day 8, Day 15 and Day 29 (FAS Set). | FAS | X |
| 14.2.20.1 | Proportion of patients with VAS pain score of "0-0.4 cm" (no eye pain) compared to placebo at Day 3, Day 8, Day 15 and Day 29 (FAS non-RM set). | FAS<br>non-<br>RM | X |
| 14.2.20.2 | Proportion of patients with VAS pain score of "0-0.4 cm" (no eye pain) compared to placebo at Day 3, Day 8, Day 15 and Day 29 (FAS Set). | FAS | X |

## 14.3 SAFETY DATA

## **Adverse events**

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.3.1.1 | Summary of Treatment Emergent Adverse Events (TEAEs) | SAF | X |
| 14.3.1.2.1 | Treatment Emergent Adverse Events by System Organ Class and Preferred Term | SAF | |
| 14.3.1.2.2 | Treatment Emergent Ocular Adverse Events by System Organ Class and Preferred Term | SAF | |
| 14.3.1.3 | TEAEs by SOC and PT by worst severity | SAF | |
| 14.3.1.4 | TEAEs by SOC and PT by worst relationship | SAF | |
| 14.3.1.5 | TEAEs related to IMP/Placebo | SAF | |
| 14.3.1.6 | TEAEs leading to discontinuation | SAF | |
| 14.3.1.7 | Serious TEAEs | SAF | |
| 14.3.1.8 | Serious TEAEs related to IMP/Placebo | SAF | |
| 14.3.1.9 | TEAEs AESI | SAF | |
| 14.3.1.10 | TEAEs AESI related to IMP/Placebo | SAF | |
| 14.3.2 | Listings of Deaths Other Serious Adverse Events, and OtherSignificant Adverse Events | SAF | |

## 14.3.3 [This title is reserved for narratives.]

Study Code: CLOBOF3-16IA01 Date: 09-JUL-2021

NCT No.: NCT04246801

Sponsor: Laboratorios Salvat, S.A.

## **Other Safety assessments**

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.3.4.1 | Absolute and Percentage change from Baseline in Vital Signs by treatment regimen. Descriptive Statistics | SAF | |
| 14.3.4.2 | Summary statistics. Change from Baseline to Day 3, Day 8, Day 15 and Day 29 compared to placebo in intraocular pressure (IOP). | SAF | X |

## **Treatment exposure**

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.3.5.1 | Compliance with IMP/Placebo % (doses/amount). Descriptive statistics. | SAF | |
| 14.3.5.2 | Exposure to IMP/Placebo: Duration of treatment Number ofdoses completed/not completed, and reasons by treatment regimen. Descriptive statistics | SAF | |

## **Concomitant medications**

| Table | Title | Pop | Top.Line |
|---|---|---|---|
| 14.3.10.1 | Summary of Prior Medications and Therapies tabulated by ATC level 3 group and generic medication name | SAF | |
| 14.3.10.2 | Summary of All Concomitant Medications (rescue and prohibited medications included) and Therapies tabulated by ATC level 3 group and generic medication name | SAF | |
| 14.3.10.3 | Summary of Concomitant Medications (Rescue and prohibited) tabulated by ATC level 3 group and generic medication name | SAF | |

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01 NCT No.: NCT04246801

# 8.2 Listings of individual patient data and other information to be produced for the clinical study report (sections 16.1 and 16.2 according to ICH E3)

| Listing | Title | Pop | Top.Line |
|---------|----------------------|-----|----------|
| 16.1.7 | Randomisation scheme | ALL | |

## Patient disposition

| Listing | Title | Pop | Top.Line |
|---|---|---|---|
| 16.2.1.1 | Patient Disposition | ALL | |
| 16.2.1.2 | Screening Failures, Discontinued Subjects, Reason for Discontinuation | ALL | X |
| 16.2.1.3 | Visits dates | | |
| 16.2.2.1 | Protocol Deviations | ALL | |
| 16.2.3.1 | Patients excluded from SAF | ALL | |
| 16.2.3.2 | Patients excluded from FAS | ALL | |
| 16.2.3.3 | Patients excluded from PP | ALL | |

# **Demographic and baseline characteristics**

| Listing | Title | Pop | Top.Line |
|---|---|---|---|
| 16.2.4.1 | Demographic data | SAF | |
| 16.2.4.2 | Relevant Medical History | SAF | |
| 16.2.4.4 | Urine Pregnancy test | SAF | |
| 16.2.4.5 | Cataract diagnosis | SAF | |
| 16.2.4.5 | Inclusion Criteria Not Met and Exclusion Criteria Met | SAF | |

## **Compliance**

| Listing | Title | Pop | Top.Line |
|---------|-----------------------------|-----|----------|
| 16.2.5 | Compliance with IMP/Placebo | SAF | |

## Efficacy data

| Listing | Title | Pop | Top.Line |
|----------|------------------------|-----|----------|
| 16.2.6.1 | Slit Slamp Examination | SAF | |
| 16.2.6.2 | BCVA by Snellen chart | SAF | |
| 16.2.6.3 | Eye pain (VAS) | SAF | |
| 16.2.6.4 | Eye discomfort | SAF | |
| 16.2.6.5 | Photophobia | SAF | |

Sponsor: Laboratorios Salvat, S.A. Study Code: CLOBOF3-16IA01

NCT No.: NCT04246801

| 16.2.6.6 | Indirect ophthalmoscopy | SAF |
|----------|-------------------------|-----|
|----------|-------------------------|-----|

## **Adverse Events**

| Listing | Title | Pop | Top.Line |
|----------|----------------|-----|----------|
| 16.2.7.1 | Adverse Events | SAF | |

## **Other Safety assessments**

| Listing | Title | Pop | Top.Line |
|-----------|--------------------------------------|-----|----------|
| 16.2.9 | Vital signs | SAF | |
| 16.2.10.1 | Physical examination | SAF | |
| 16.2.10.2 | Eye examination | SAF | |
| 16.2.11 | IOP measurementsby Goldman Tonometer | SAF | |

# **Concomitant medication**

| Listing | Title | Pop | Top.Line |
|---|---|---|---|
| 16.2.12.1 | Prior Medications and Therapies tabulated by ATC level 3 group and WHO preferred name | SAF | |
| 16.2.12.2 | All Concomitant Medications and Therapies tabulated by ATC level 3 group and WHO preferred name | SAF | |
| 16.2.12.3 | Rescue and prohibited Concomitant Medications tabulated by ATC level 3 group and WHO preferred name | SAF | |